CLINICAL TRIAL: NCT01532544
Title: Double-blinded, Randomized Trial in Severe Pneumonia Patients With Severe Sepsis Investigating the Safety and Efficacy of Co-administration of Iloprost and Ascending Doses of Eptifibatide Compared to Low-molecular-weight Heparin
Brief Title: Integrilin and Ilomedin in Combination in Comparison to Standard Treatment in Severe Pneumonia Patients With Severe Sepsis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting patients, company closed down
Sponsor: Thrombologic ApS (Industry)
Collaborators: Anders Perner (Unknown); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-PS-03; 2011-002254-31 (EudraCT Number)
Record Dates: First submitted 2012-01-30; First posted 2012-02-14 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Pneumonia
Keywords: Severe pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Eptifibatide; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrilin and Ilomedin given as continous infusion (Experimental)
  Interventions: Drug: Ilomedin and Integrilin
- Standard treatment daily doses of low molecular weight heparin (Placebo Comparator): Standard treatment daily doses of low molecular weight heparin.
  Interventions: Drug: low molecular weight heparin.

INTERVENTIONS:
Drug: Ilomedin and Integrilin — Continuous infusion
  Other Names: Integrilin and Ilomedin
  Arms: Integrilin and Ilomedin given as continous infusion
Drug: low molecular weight heparin.
  Arms: Standard treatment daily doses of low molecular weight heparin

SUMMARY:
This is an investigator sponsored double-blinded, multinational, multi center, randomized (2:1 active:placebo), placebo-controlled, phase IIa trial in severe pneumonia patients with severe sepsis or septic shock, investigating the safety and efficacy of co-administration of Iloprost and escalating doses of Eptifibatide for continuous intravenous infusion in totally 36 patients.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age AND
2. Suspected or proven bacterial pneumonia requiring administration of antibiotics:

   * Clinical diagnosis of pneumonia, (i.e. new or increased cough, production of purulent sputum or a change in the character of sputum in subjects who normally have purulent sputum, typical auscultatory findings of pneumonia on chest examination) and:
   * chest radiograph or CT within the last 24 hr showing a pulmonary infiltrate.
3. Dyspnea and/or tachypnea (>20 breaths/minute) or mechanical ventilation
4. Two or more systemic inflammatory response syndrome (SIRS) criteria within the last 24 hours:

   * Temperature </= 36˚ C or >/= 38˚C
   * Heart rate >/= 90 beats per minute
   * Mechanical ventilation for acute respiratory process or respiratory rate >/= 20 breaths per minute or PaC02 < 4.2 kPa
   * WBC >/= 12,000/mm³ OR </= 4,000/mm³ OR > 10% bands
5. At least one organ failure beyond respiratory failure (cerebral, cardiovascular, hepatic, renal or coagulation within the last 24 hours (> 2 in SOFA score for the specific organ system) AND
6. Can be randomized into trial and dosed < 48 h after severe sepsis diagnosis AND
7. Consent is obtainable -

Exclusion Criteria:

1. Patient is pregnant or breast-feeding
2. Patient weigh more than 125 kg
3. Patients with known allergy towards any of the investigational products or contraindications which should be excluded according to the investigational product specifications
4. Investigators clinical decision deeming study participation not favourable for the patient
5. Patients in whom the clinician finds antithrombotic therapy contraindicated - prophylaxis included
6. Patients at increased risk of bleeding: Surgery in the previous 12 h, expected surgery within 72 h, epidural or spinal puncture in the previous 12 h, platelet count less than 30,000/mm3 in the previous 24 h, INR above 2.0 in the previous 24 h, need of blood products for bleeding in the previous 24 h, treatment with any antithrombotics within 12 h (profylaxis excepted), current or previous intracranial bleeding or traumatic brain or spinal injury within the last month.
7. Patients requiring any form of antithrombotics (beyond profylaxis) in therapeutic doses or prothrombotics in any dose, including,

   * unfractionated heparin within 8 hours before the infusion (prophylactic heparin up to 15,000 U/day permitted).
   * Low-molecular-weight heparin within 12 hours (prophylactic doses permitted).
   * exceeded the upper limit of normal.
   * Acetylsalicylic acid more than 650 mg/day within 3 days before the study.
   * Thrombolytic therapy within 3 days before the study (catheter clearance doses permitted).
   * Glycoprotein IIb-IIIa antagonists within 7 days before the study.
   * Antithrombin III with dose greater than 10,000 U within 12 hours before the study.
   * Protein C within 24 hours of the study.
8. Previous diagnosed condition that might mimic or complicate the course and evaluation of the infectious disease process (severe bronchiectasis, lung abcess or empyema, aspiration pneumonia, active tuberculosis, pulmonary malignancy, cystic fibrosis, severe chronic interstitial pneumonia, COPD or other forms of chronic lung disease requiring home oxygen treatment or resulting in chronic CO2 retention, , etc.)
9. Patient not expected to survive more than 30 days because of uncorrectable medical or surgical condition other than sepsis
10. Patient with acute or chronic renal failure requiring dialysis (renal failure without need for dialysis permitted).
11. Patient with hematological malignancies of any kind
12. Patients who have undergone transplantation of bone marrow, liver, pancreas, heart, lung, or bowel (kidney transplant permitted)
13. Patient has known hypercoagulable condition:

    APC resistance Hereditary protein C, protein S, or antithrombin III deficiency Anticardiolipin or antiphospholipid antibody Lupus anticoagulant Homocysteinemia Recent or highly suspected pulmonary embolism or deep venous thrombosis (within 3 months)
14. Patients with known congenital hypocoagulable diseases
15. Patient with known AIDS
16. Patient with known primary pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in platelet count from baseline to 72 hours post treatment | 11 bloodsamples over 7 days
  Will be from pre-study drug administration until 7 days

SECONDARY OUTCOMES:
Severe bleeding (intracranial or clinical bleeding with the use of 3 RBC units or more) (KyperSept trial) | 7 days
  If longer in the ICU ward followed until discharged.
Days of vasopressor, ventilator and renal replacement therapy and use of blood product (in ICU) after randomization | 7 days
  Followed longer if not discharged from the ICU at day 7

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (2):
  - University hospital Copenhagen, Copenhagen
  - Vejle hospital, Vejle
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: Undecided